CLINICAL TRIAL: NCT07136961
Title: Efficacy and Safety of Robotic-assisted Bronchoscopy Combined With the ICNVA Strategy in Biopsy of Peripheral Pulmonary Nodules: A Prospective, Single-center, Single-arm Study
Brief Title: Efficacy and Safety of Robotic-assisted Bronchoscopy Combined With the ICNVA Strategy in Biopsy of Peripheral Pulmonary Nodules
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Shaohua Dai, M.D., Ph.D, Professor, The First Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSH1
Record Dates: First submitted 2025-08-09; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lung Nodules; Biopsy; Navigation, Spatial
Keywords: bronchial navigation and positioning
MeSH Terms: conditions — Spatial Navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-Assisted Bronchoscopy (RAB) (Experimental): 1. Preoxygenation & Navigation Registration
  2. Robotic-Guided Navigation
  3. Puncture Tunnel Establishment
  4. Position Verification & Adjustment
     Perform confirmatory CT scan to assess tool-nodule relationship:
     Tool-in-lesion (TIL) : Biopsy tool penetrates nodule Center Strike : Tool tip reaches central 1/3 of nodule (coronal/sagittal/horizontal planes) Tool-touch-lesion : Tool contacts but does not enter nodule
     * 4mm deviation : Proceed to biopsy >4mm deviation : Adjust based on operator judgment
  5. Biopsy & Rapid Evaluation Obtain tissue samples Conduct ROSE (Rapid On-Site Evaluation) to guide next steps
  6. Post-Procedure Safety Check Perform postoperative CT to exclude pneumothorax/hemorrhage Maintain identical ventilation settings during imaging and biopsy phases to prevent target shift
  Interventions: Procedure: Robot-Assisted Bronchoscopy (RAB)

INTERVENTIONS:
Procedure: Robot-Assisted Bronchoscopy (RAB) — 1. Preoxygenation & Navigation Registration
  2. Robotic-Guided Navigation
  3. Puncture Tunnel Establishment
  4. Position Verification & Adjustment
     Perform confirmatory CT scan to assess tool-nodule relationship:
     Tool-in-lesion (TIL) : Biopsy tool penetrates nodule Center Strike : Tool tip reaches central 1/3 of nodule (coronal/sagittal/horizontal planes) Tool-touch-lesion : Tool contacts but does not enter nodule
     * 4mm deviation : Proceed to biopsy >4mm deviation : Adjust based on operator judgment
  5. Biopsy & Rapid Evaluation Obtain tissue samples Conduct ROSE (Rapid On-Site Evaluation) to guide next steps
  6. Post-Procedure Safety Check Perform postoperative CT to exclude pneumothorax/hemorrhage Maintain identical ventilation settings during imaging and biopsy phases to prevent target shift

SUMMARY:
To assess the efficacy and safety of robotic-assisted bronchoscopy system (bronchial navigation and positioning device) combined with ICNVA strategy for peripheral pulmonary nodule biopsy through a prospective, single-center, single-arm study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, and ≤75 years old, male or female;
2. Patients with peripheral lung lesions found by chest CT, whose diameter ≥ 6mm and < 3cm, who plan to undergo robotic-assisted bronchoscopic for pulmonary biopsy;
3. The patient voluntarily undergo bronchoscopy and meet the requirements for bronchoscopy;
4. Patients can understand the purpose of the trial, have good compliance with the examination and follow-up, voluntarily participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

1. Patients with cardiovascular diseases, such as blood pressure instability, myocardial infarction or arrhythmia;
2. Patients with massive hemoptysis within two weeks;
3. Patients with severe pneumothorax and rib fracture;
4. Patients with serious infectious diseases, such as tuberculosis or AIDS;
5. Patients with severe abdominal aortic aneurysm or thoracic aortic aneurysm;
6. Participants who have participated in or are participating in drug clinical trials within 3 months before screening, or have participated in other medical device clinical trials within 30 days;
7. Those who were not considered suitable for inclusion by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Tool-in-lesion rate | Perioperative/Periprocedural

SECONDARY OUTCOMES:
Center Strike rate | Perioperative/Periprocedural
Tool-touch-lesion rate | Perioperative/Periprocedural
Successful diagnosis rate | Perioperative/Periprocedural
Lesion detection rate | Perioperative/Periprocedural
Bronchopulmonary hemorrhage rate | Perioperative/Periprocedural
Pneumothorax rate | Perioperative/Periprocedural
CT to Body divergence（CTBD） | Perioperative/Periprocedural
  The difference between the distance from the probe to the center of the target nodule in Robotic-Assisted Bronchoscopy and the actual distance from the probe to the target nodule center in follow-up Computed Tomography
Successful operation rate | Perioperative/Periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No